CLINICAL TRIAL: NCT02348086
Title: Autologous Adipose Stromal Vascular Fraction Outcomes in Rheumatoid Arthritis Research Study
Brief Title: Outcomes Data of Adipose Stem Cells to Treat Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: StemGenex (Industry)
Responsible Party: Sponsor
Other Study IDs: SVF01RA; ASCRA-01 (Other: StemGenex)
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the impact that treatment with a cellular concentrate derived from an individual's own fat, known as the stromal vascular fraction (SVF), has on pain and functionality in people with rheumatoid arthritis (RA). SVF contains multiple cellular components, including stem cells, with both regenerative and anti-inflammatory properties. This therapy has shown promise for ameliorating the symptoms of RA. This study is designed to evaluate changes in pain and functionality in individuals with RA for up to 12 months following SVF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with rheumatoid arthritis
* Subjects scheduled for a stem cell/SVF treatment
* Subjects willing and able to sign informed consent
* Subjects willing and able to perform follow-up interviews and surveys

Exclusion Criteria:

* Subjects with addition major health condition/disease diagnoses
* Subjects that are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Overall Rheumatoid Arthritis Disease Activity Over the Course of a 12 Month Period as Measured by the Patient Activity Scale-II (PAS-II) | Baseline, 12 Months
  The change from baseline over the course of 12 months using participants' assessment of their overall ability to be active. Mean scores will be used for baseline (day 0) and all interviews up to month 12 (months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12). Answer options are graded either according to a four point or ten point Likert response scale.

SECONDARY OUTCOMES:
Change from Baseline in Overall Health at Month 12 as Measured by the Participants' Response to the Health Assessment Questionnaire-II (HAQ-II) | Baseline, Month 12
  Participant assessment of the change in their overall health from baseline to month 12 using the HAQ-II. Answer options are given as a four point Likert response scale.
Change from Baseline in Overall Pain at Month 12 as Measured by Participants' Response to the Patient Activity Scale-II (PAS-II) Pain Subscale | Baseline, Month 12
  Participant assessment of the change in their overall pain from baseline to month 12 using the PAS-II pain subscale. Answer options are given as a ten point Likert response scale.
Change from Baseline in Overall Global Activity at Month 12 as Measured by Participants' Response to the Patient Activity Scale-II (PAS-II) Global Activity Subscale | Baseline, Month 12
  Participant assessment of the change in their overall global activity from baseline to month 12 using the PAS-II global activity subscale. Answer options are given as a ten point Likert response scale.

CONTACTS AND LOCATIONS:
Locations (1):
- StemGenex, San Diego, California, United States